CLINICAL TRIAL: NCT04755387
Title: EASTYLE (DE-escAlation Strategy for Optimal Ticagrelor Therapy in Acute MYocardiaL Infarction PatiEnts, Prospective, Multicenter, Randomized) Trial
Brief Title: Ticagrelor De-escalation Strategy in AMI Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A University (Other)
Collaborators: Biotronik SE & Co. KG (Industry); Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Moo Hyun Kim, Professor, Deptartment of Cardiology, Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASTYLE
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Ticagrelor; DAPT; De-escalation strategy; Abbreviated strategy
MeSH Terms: interventions — Ticagrelor; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- De-escalation strategy (Experimental): PCI ~ 1 month: ticagrelor 90 mg twice daily + aspirin 100 mg once daily
  1 ~ 3 months: ticagrelor 60 mg twice daily + aspirin 100 mg once daily
  3 ~ 12 months: ticagrelor 60 mg twice daily
  Interventions: Drug: De-escalation strategy
- Conventional strategy (Active Comparator): PCI ~ 12 months: ticagrelor 90 mg twice daily + aspirin 100 mg once daily
  Interventions: Drug: Conventional strategy

INTERVENTIONS:
Drug: De-escalation strategy — De-escalation strategy indicates conventional DAPT (ticagrelor 90 mg twice daily + aspirin 100 mg once daily) for 1 month, followed by de-escalation DAPT (ticagrelor 60 mg twice daily + aspirin 100 mg once daily) between 1 and 3 months. Between 3 and 12 months, patients will be treated with ticagrelor monotherapy (ticagrelor 60 mg twice daily).
  Other Names: Ticagrelor 60 mg, aspirin early discontinuation
  Arms: De-escalation strategy
Drug: Conventional strategy — Conventional stratetgy indicates conventional DAPT including ticagrelor 90 mg twice daily and aspirin 100 mg once daily during 12 months.
  Other Names: Ticagrelor 90 mg, DAPT
  Arms: Conventional strategy

SUMMARY:
DAPT de-escalation strategies to reduce bleeding include de-escalation of DAPT intensity (downgrading from potent P2Y12 inhibitor at conventional doses to either clopidogrel or reduced-dose prasugrel) or abbreviation of DAPT duration. The EASTYLE trial will evaluate a hybrid DAPT de-escalation strategy (reduced-dose ticagrelor, followed by aspirin early discontinuation) in AMI patients, compared with a conventional DAPT strategy.

DETAILED DESCRIPTION:
In ACS patients undergoing percutaneous coronary intervention, conventional dual antiplatelet therapy (DAPT) for patients with acute coronary syndromes undergoing percutaneous coronary intervention comprises aspirin with a potent P2Y12 inhibitor (prasugrel or ticagrelor) for 12 months. Although this approach reduces ischaemic risk, patients are exposed to a substantial risk of bleeding during the stabilized period. Strategies to reduce bleeding include de-escalation of DAPT intensity (downgrading from potent P2Y12 inhibitor at conventional doses to either clopidogrel or reduced-dose prasugrel) or abbreviation of DAPT duration. Abbreviation of DAPT duration after 1-6 months, followed by monotherapy with aspirin or a P2Y12 inhibitor, reduces bleeding without an increase in ischaemic events in patients at high bleeding risk, particularly those without high ischaemic risk. Either strategy requires assessment of the ischaemic and bleeding risks of each individual. Previous clinical and laboratory evidence demonstrates that a conventional-dose of ticagrelor has a potent antiplatelet effect, which appears to have a potential to increase the risk of bleeding during the stabilized period. Adjunctive use of aspirin to P2Y12 inhibitor would be important to protect the risk of thrombotic events in AMI patients, which use has a limited benefit with increased bleeding rate during the the stabilized period.

The EASTYLE trial will evaluate clinical benefit of step-down de-escalation DAPT strategy including downgrading of P2Y12 inhibition (from 90 mg to 60 mg ticagrelor at 1 month post-PCI) and abbreviation of DAPT duration (aspirin discontinuation at 3 months post-PCI), compared with a conventional DAPT strategy in AMI patients. This trial will support that the optimal platelet inhibition would be attenuated over time even in AMI patients. The result will make a big step toward precision medicine in the field of antiplatelet treatment in AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with acute myocardial infarction.
* Age ≥19 year-old
* Successful PCI with ultrathin bioresorbable polymer sirolimus-eluting stents (Orsiro; Biotronik AG).
* Provision of informed consent.

Exclusion Criteria:

* Any prior event of hemorrhagic stroke or ICH.
* Active bleeding (e.g., GI bleeding, ICH) or high-risk of serious bleeding.
* Bleeding diathesis or coagulopathy (e.g., hemoglobin ≤ 10 g/dL or platelet count < 100,000/μL, bleeding needing transfusion within 30 days, and so on).
* Allergy to stent metal, contrat media, and antiplatelet regimens.
* Moderate to severe hepatic dysfunction (Child-Pugh class B or C).
* Need for oral anticoagulation therapy.
* Current or potential pregnancy.
* Currently treated with strong CYP3A4 inhibitors.
* Life expectancy <1 year.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2312 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint (NACE) | 12 months
  MACCE (all-cause death, non-fatal myocardial infarction, stent thrombosis or non-fatal stroke) + major bleeding (BARC type 2, 3, or 5 bleeding)

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  all-cause death, non-fatal myocardial infarction, stent thrombosis or non-fatal stroke
Bleeding events | 12 months
  BARC type 2, 3 or 5 bleeding; BARC 3 or 5 bleeding; TIMI major or minor bleeding; GUSTO severe or moderate bleeding; ISTH major bleeding
All-cause death | 12 months
  any mortality
CV death | 12 months
  Death related CV system
MI | 12 months
  Myocardial infarction
Stent thrombosis | 12 months
  definite or probable stent thrombosis by Academic Research Consortium (ARC) definition
Ischemic stroke | 12 months
  Stroke
Cardiac death, or MI | 12 months
  Coronary thrombotic events
Cardiac death, MI or stent thrombosis | 12 months
  Coronary thrombotic events
Cardiovascular death, MI or stroke | 12 months
  MACE
TLR | 12 months
  target lesion revascularization
TVR | 12 months
  target vessel revascularization
Any revascularization | 12 months
  Re-PCI during follow-up

OTHER OUTCOMES:
Type of AMI | 12 months
  STEMI vs. NSTEMI
HBR | 12 months
  presence of HBR (high bleeding risk) criteria
DM | 12 months
  presence of diabetes mellitus
CKD | 12 months
  presence of chronic kidney disease
Anemia | 12 months
  presence of anemia
Gender | 12 months
  Male vs. female
Age | 12 months
  Old vs. young age (65 yo, 75 yo)
Complex PCI | 12 months
  Presence of complex PCI
GDMT | 12 months
  Presence of guideline-directed medical therapy
Type of statin | 12 months
  Rosuvastatin vs. other statins
CHF | 12 months
  Presence of congestive heart failure
PAD | 12 months
  Presence of peripheral artery disease
PFT | 12 months
  VerifyNow assy
Predictors of MACCE | 12 months
  Clinical impact of de-esclation strategy on MACCE
Predictors of maor bleeding | 12 months
  Clinical impact of de-esclation strategy on major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, PhD, Principal Investigator — Dong-A University Hospital, Busan, Republic of Korea
Locations (1):
- DongA University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goto S, Huang CH, Park SJ, Emanuelsson H, Kimura T. Ticagrelor vs. clopidogrel in Japanese, Korean and Taiwanese patients with acute coronary syndrome -- randomized, double-blind, phase III PHILO study. Circ J. 2015;79(11):2452-60. doi: 10.1253/circj.CJ-15-0112. Epub 2015 Sep 16. PMID 26376600
- [Background] Jin C, Kim MH, Bang J, Serebruany V. A Prospective, Randomized, Open-Label, Blinded, Endpoint Study Exploring Platelet Response to Half-Dose Prasugrel and Ticagrelor in Patients with the Acute Coronary Syndrome: HOPE-TAILOR Study. Cardiology. 2017;138(4):201-206. doi: 10.1159/000478000. Epub 2017 Aug 16. PMID 28810251
- [Background] Gorog DA, Ferreiro JL, Ahrens I, Ako J, Geisler T, Halvorsen S, Huber K, Jeong YH, Navarese EP, Rubboli A, Sibbing D, Siller-Matula JM, Storey RF, Tan JWC, Ten Berg JM, Valgimigli M, Vandenbriele C, Lip GYH. De-escalation or abbreviation of dual antiplatelet therapy in acute coronary syndromes and percutaneous coronary intervention: a Consensus Statement from an international expert panel on coronary thrombosis. Nat Rev Cardiol. 2023 Dec;20(12):830-844. doi: 10.1038/s41569-023-00901-2. Epub 2023 Jul 20. PMID 37474795
- [Background] Gorog DA, Jeyalan V, Markides RIL, Navarese EP, Jeong YH, Farag M. Comparison of De-escalation of DAPT Intensity or Duration in East Asian and Western Patients with ACS Undergoing PCI: A Systematic Review and Meta-analysis. Thromb Haemost. 2023 Aug;123(8):773-792. doi: 10.1055/s-0043-57030. Epub 2023 Apr 18. PMID 37072035
- [Background] Kang MG, Ahn JH, Kim K, Koh JS, Park JR, Hwang SJ, Park Y, Tantry US, Gurbel PA, Hwang JY, Jeong YH. Prevalence of adverse events during ticagrelor versus clopidogrel treatment and its association with premature discontinuation of dual antiplatelet therapy in East Asian patients with acute coronary syndrome. Front Cardiovasc Med. 2022 Dec 12;9:1053867. doi: 10.3389/fcvm.2022.1053867. eCollection 2022. PMID 36578832
- [Background] Kubica J, Adamski P, Gorog DA, Kubica A, Jilma B, Budaj A, Siller-Matula JM, Gurbel PA, Alexopoulos D, Badariene J, Dabrowski P, Dudek D, Giannitsis E, Horszczaruk G, Jaguszewski MJ, James S, Jeong YH, Kryjak M, Niezgoda P, Ostrowska M, Patti G, Romanek J, Di Somma S, Specchia G, Tantry U, Gasior M, Tycinska A, Wojakowski W, Buszko K, Gil R, Gruchala M, Kasprzak J, Kleinrok A, Legutko J, Lesiak M, Navarese EP. Low-dose ticagrelor with or without acetylsalicylic acid in patients with acute coronary syndrome: Rationale and design of the ELECTRA-SIRIO 2 trial. Cardiol J. 2022;29(1):148-153. doi: 10.5603/CJ.a2021.0118. Epub 2021 Oct 8. No abstract available. PMID 34622433
- [Background] Kim L, Choe JC, Ahn JH, Lee HW, Oh JH, Choi JH, Lee HC, Cha KS, Hong TJ, Jeong YH, Park JS. Temporal Trends of Bleeding Episodes during Half- vs. Standard-Dose Ticagrelor in Acute Coronary Syndrome Patients with Low Platelet Reactivity: A Randomized BLEEDING-ACS Trial. J Clin Med. 2021 Mar 10;10(6):1159. doi: 10.3390/jcm10061159. PMID 33802015
- [Background] Kim HK, Tantry US, Smith SC Jr, Jeong MH, Park SJ, Kim MH, Lim DS, Shin ES, Park DW, Huo Y, Chen SL, Bo Z, Goto S, Kimura T, Yasuda S, Chen WJ, Chan M, Aradi D, Geisler T, Gorog DA, Sibbing D, Lip GYH, Angiolillo DJ, Gurbel PA, Jeong YH. The East Asian Paradox: An Updated Position Statement on the Challenges to the Current Antithrombotic Strategy in Patients with Cardiovascular Disease. Thromb Haemost. 2021 Apr;121(4):422-432. doi: 10.1055/s-0040-1718729. Epub 2020 Nov 10. PMID 33171520
- [Background] Park Y, Koh JS, Lee JH, Park JH, Shin ES, Oh JH, Chun W, Lee SY, Bae JW, Kim JS, Kim W, Suh JW, Yang DH, Hong YJ, Chan MY, Kang MG, Park HW, Hwang SJ, Hwang JY, Ahn JH, Choi SW, Jeong YH; HEALING-AMI Investigators. Effect of Ticagrelor on Left Ventricular Remodeling in Patients With ST-Segment Elevation Myocardial Infarction (HEALING-AMI). JACC Cardiovasc Interv. 2020 Oct 12;13(19):2220-2234. doi: 10.1016/j.jcin.2020.08.007. PMID 33032710